CLINICAL TRIAL: NCT06082596
Title: A Multicenter, Open, Phase I Clinical Study of BEBT-908 for Injection in the Treatment of Relapsed Refractory Malignant Lymphoma, Multiple Myeloma and Chronic Lymphoblastic Leukemia
Brief Title: Study of BEBT-908 in Subjects With Advanced Hematological Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeBetter Med Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBMT-908-P01
Record Dates: First submitted 2023-10-09; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Relapsed or Refractory Non-Hodgkin's Lymphoma; Relapsed or Refractory Multiple Myeloma
Keywords: BEBT-908 for injection; Safety; Tolerability; Pharmacokinetics; Effectiveness
MeSH Terms: conditions — Recurrence; Lymphoma, Non-Hodgkin; Multiple Myeloma | interventions — BEBT-908; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Monotherapy group 1(Dose escalation phase) (Experimental): BEBT-908 for injection， dosage form ：Injection； specification: 25 mg , administration method: 10mg/m2，intravenous drip, firstly the subjects were given a single dose and observed for 6 days. At the end of the observation period, if the subjects were tolerant to a single dose and safe, they would receive the same dose for a cycle (21 days), giving the drug three times a week for 2 weeks and stopping the drug for 1 week. A total of 21 days is a cycle.
  Interventions: Drug: BEBT-908 for injection
- Monotherapy group 2(Dose escalation phase) (Experimental): BEBT-908 for injection， dosage form ：Injection； specification: 25 mg , administration method: 15mg/m2，intravenous drip, firstly the subjects were given a single dose and observed for 6 days. At the end of the observation period, if the subjects were tolerant to a single dose and safe, they would receive the same dose for a cycle (21 days), giving the drug three times a week for 2 weeks and stopping the drug for 1 week. A total of 21 days is a cycle.
  Interventions: Drug: BEBT-908 for injection
- Monotherapy group 3(Dose escalation phase) (Experimental): BEBT-908 for injection， dosage form ：Injection； specification: 25 mg , administration method: 22.5mg/m2，intravenous drip, firstly the subjects were given a single dose and observed for 6 days. At the end of the observation period, if the subjects were tolerant to a single dose and safe, they would receive the same dose for a cycle (21 days), giving the drug three times a week for 2 weeks and stopping the drug for 1 week. A total of 21 days is a cycle.
  Interventions: Drug: BEBT-908 for injection
- Monotherapy group 4(Dose escalation phase) (Experimental): BEBT-908 for injection， dosage form ：Injection； specification: 25 mg , administration method: 33.75mg/m2，intravenous drip, firstly the subjects were given a single dose and observed for 6 days. At the end of the observation period, if the subjects were tolerant to a single dose and safe, they would receive the same dose for a cycle (21 days), giving the drug three times a week for 2 weeks and stopping the drug for 1 week. A total of 21 days is a cycle.
  Interventions: Drug: BEBT-908 for injection
- Monotherapy group 5(Dose escalation phase) (Experimental): BEBT-908 for injection， dosage form ：Injection； specification: 25 mg , administration method: 45mg/m2，intravenous drip, firstly the subjects were given a single dose and observed for 6 days. At the end of the observation period, if the subjects were tolerant to a single dose and safe, they would receive the same dose for a cycle (21 days), giving the drug three times a week for 2 weeks and stopping the drug for 1 week. A total of 21 days is a cycle.
  Interventions: Drug: BEBT-908 for injection
- Monotherapy group 6（Dose expansion phase） (Experimental): BEBT-908 for injection ，dosage form ：Injection ；specification: 25mg , administration method: 15mg/m2，intravenous drip, 3 times a week, continuous administration for 2 weeks and withdrawal for 1 week，21 days as cycle, until the disease progressed or withdrew.
  Interventions: Drug: BEBT-908 for injection
- Monotherapy group 7（Dose expansion phase） (Experimental): BEBT-908 for injection ，dosage form ：Injection ；specification: 25mg , administration method: 22.5mg/m2，intravenous drip, 3 times a week, continuous administration for 2 weeks and withdrawal for 1 week，21 days as cycle, until the disease progressed or withdrew.
  Interventions: Drug: BEBT-908 for injection

INTERVENTIONS:
Drug: BEBT-908 for injection — Dose escalation phase：10 or 15、22.5、33.75、45mg/m2, intravenous drip, firstly single dose, after the observation period, the drug was administered continuously for 1 cycle (21 days), 3 times a week, continuous administration for 2 weeks and withdrawal for 1 week.
  Dose expansion phase：15 or 22.5mg/m2，intravenous drip, 3 times a week, continuous administration for 2 weeks and withdrawal for 1 week，21 days as cycle.
  Other Names: CUDC-908

SUMMARY:
The purpose of this study was to evaluate the safety and tolerance of BEBT-908 for injection in the treatment of recurrent refractory malignant lymphoma, multiple myeloma and chronic lymphoblastic leukemia, and to obtain the pharmacokinetic data and preliminary efficacy of BEBT-908 for injection, and to explore the relationship between the safety and efficacy of BEBT-908 for injection and related biomarkers.

DETAILED DESCRIPTION:
This study is divided into two stages: dose increasing stage and expanding into the group.

Dose escalation phase: The initial dose was 10mg/m2, and the subsequent dose group was increased by 100% until the first case of grade 2 non-blood toxicity or grade 3 hematological toxicity related to the test drug and no dose-limiting toxicity, then the dose was increased by 50%, and a total of 5 dose groups were designed. In this stage, all subjects received a single dose first and were observed for 6 days. After the end of the observation period, if the subjects were safely tolerant to a single dose，then will receive the same dose of treatment for a cycle, administration regimen is 3 times a week, continuous administration for 2 weeks, withdrawal for 1 week, a total of 21 days as a cycle.

Dose expansion phase: according to the results of pharmacokinetics, safety and efficacy of BEBT-908 for injection obtained in the dose escalation phase, we plan to select two doses to further observe the safety, pharmacokinetic characteristics and preliminary efficacy of BEBT-908 for injection in about 20-40 subjects with non-Hodgkin's malignant lymphoma. In this stage, all dose groups were administered continuously for 2 weeks and stopped for 1 week for a total of 21 days，until the disease progresses or withdraws.

Participants will need to understand the requirements and risks of the trial, sign an informed consent form, accept the dosing regimen required by the trial protocol, and follow the investigator's guidance.

ELIGIBILITY:
Inclusion Criteria:

* Dose escalation phase:

  1. Age ≥ 18 and ≤ 70 years old, both men and women.
  2. Tissue biopsy, bone marrow examination and / or hematological examination confirmed relapsed refractory （Note 1） malignant lymphoma, chronic lymphoblastic leukemia and multiple myeloma. （Note 2 and Note 3）
  3. With measurable lesions . (Note 4)
  4. Eastern Cooperative Oncology Group (ECOG) score≤2.
  5. The level of organ function must meet the following requirements:

Bone marrow:

1. Absolute neutrophil count (ANC) ≥ 1000 /μL (if recent bone marrow biopsies or smears prove tumor progression, this index can be < 1000/μL).
2. Hemoglobin (HGB) ≥ 9g/dL.
3. Platelet count (PLT) ≥ 1000000/μL (if recent bone marrow biopsies or smears prove tumor progression, this index can be < 1000000/μL).

Liver function:

In patients with serum bilirubin ≤ 1.5 ×upper limit of normal value (ULN) or Gilbert syndrome, the total bilirubin is less than 3.0 × ULN and direct bilirubin is within the normal range.

Serum creatinine < 1.5×ULN; Alanine aminotransferase (ALT), Aspartate aminotransferase (AST)or Alkaline phosphatase (ALP) ≤ 2.5 ×ULN.

When there is liver metastasis, ALT, AST or ALP ≤ 5 × ULN.

6.Non-pregnant women and male and female subjects who did not consider fertility during and after the trial, or who had preserved sperm or eggs in vitro before the trial, or reconsidered fertility according to reproductive function 5 years after the end of the trial.

7.After a comprehensive understanding, the subjects were willing to sign the informed consent form.

Note 1: relapse or refractory is defined as follows:

Chronic Lymphoblastic Leukemia: subjects who are ineffective after at least 2 chemotherapy regimens, and the subjects are not suitable or refuse to transplant. Relapse: the patient reached Complete Response (CR) or Partial Response (PR), and Progressive Disease (PD) ≥ 6 months later. Refractory: failed treatment (without CR or PR) or PD less than 6 months after the last chemotherapy.

Malignant Lymphoma: refractory or relapse after at least 2 chemotherapy regimens.

Multiple Myeloma: relapse or refractory is defined as relapse or disease progression after at least 2 chemotherapy regimens (refractory occurred during the last chemotherapy or within 60 days after the last medication).

Note 2: Malignant Lymphoma includes B-cell non-Hodgkin's lymphoma, B-cell Hodgkin's lymphoma, diffuse large B-cell lymphoma, T-cell lymphoma and so on.

Note 3: If the subjects can provide test results to confirm the nature of the disease and the researchers determine that the nature of the disease has not changed, there is no need for reexamination.

Note 4: For subjects with malignant lymphoma, the lesions are measured by computed tomography (CT) or magnetic resonance imaging (MRI) or positron emission tomography (PET) / PET-CT. Bone marrow biopsy or smear may be performed in the evaluation of curative effect.

For subjects with multiple myeloma, it can be accepted that bone marrow biopsy or smear may be performed during the evaluation of the curative effect.

For subjects with chronic lymphoblastic leukemia, it can be accepted that bone marrow biopsy or smear may be performed during the evaluation of the curative effect.

* Dose expansion phase:

  1. After a comprehensive understanding, the subjects were willing to sign the informed consent form.
  2. Age ≥ 18 and ≤ 70 years old, both men and women.
  3. Tissue biopsy confirmed as relapse or refractory (Note 1) non-Hodgkin's lymphoma.
  4. With measurable lesions .(Note 4)
  5. Eastern Cooperative Oncology Group (ECOG) score≤2.
  6. The level of organ function must meet the following requirements:

Bone marrow:

1. Absolute neutrophil count (ANC) ≥ 1000 /μL.
2. Hemoglobin (HGB) ≥ 8g/dL.
3. Platelet count (PLT) ≥ 1000000/μL (if recent bone marrow biopsies or smears prove tumor progression, this index can be < 1000000/μL).

Liver function:

In patients with serum bilirubin ≤ 1.5 ×upper limit of normal value (ULN) or Gilbert syndrome, the total bilirubin is less than 3.0 × ULN and direct bilirubin is within the normal range.

Serum creatinine < 1.5×ULN; Alanine aminotransferase (ALT), Aspartate aminotransferase (AST) or Alkaline phosphatase (ALP) ≤ 2.5 ×ULN.

When there is liver metastasis, ALT, AST or ALP ≤ 5 × ULN.

7.Non-pregnant women and male and female subjects who did not consider fertility during and after the trial, or who had preserved sperm or eggs in vitro before the trial, or reconsidered fertility according to reproductive function 5 years after the end of the trial.

Note 1: relapse or refractory is defined as refractory or relapse after at least 2 chemotherapy regimens.

Note 2: The lesions are measured by computed tomography (CT) or magnetic resonance imaging (MRI) or positron emission tomography (PET) / PET-CT. Bone marrow biopsy or smear may be performed in the evaluation of curative effect.

Exclusion Criteria:

* Dose escalation phase:

  1. Severe allergies to research drugs or any of their excipients are known.
  2. Because the research drugs may have genotoxicity, mutagenicity and teratogenicity, the following subjects should be excluded: men and women who plan to reproduce within 5 years without in vitro preservation of sperm or eggs before the trial, unless follow-up studies confirm reproductive safety; pregnant or lactating women.
  3. The treatment of the subjects before the trial:

     1. Bone marrow transplantation was performed within 3 months before enrolling the group.
     2. Received bone marrow inhibitory chemotherapy or biotherapy within 3 weeks before enrolling the group.
     3. Before enrolling the group, the subjects had been treated with any persistent or intermittent small molecular targeted drugs (Phosphoinositide 3-kinase (PI3K) inhibitors or Mammalian Target of Rapamycin (mTOR) inhibitors or Histone Deacetylase (HDAC) inhibitors). Subjects in the dose increasing phase of this study will not be subject to the exclusion criteria of this article if they participate in the expanded group phase screening.
     4. Within 3 months before enrolling the group, subjects received radiotherapy that affected the efficacy evaluation of this study, or local supportive radiotherapy that affected the bone marrow function of the subjects.
     5. Subjects received any hematopoietic colony stimulating factor therapy (such as granulocyte colony stimulating factor （G-CSF）, granulocyte macrophage colony stimulating factor（GM-CSF）) within 2 weeks before enrolling the group (Note 1).
     6. Major surgery was performed within 14 days before enrolling the group, or the side effects of the operation were not stable.
     7. Subjects received glucocorticoid prednisone daily >10mg (or equivalent drug) treatment within 7 days before enrollment. (Note 2)
  4. After the previous treatment (chemotherapy or biotherapy), there was persistent toxicity of grade 2 or above, which was not stable at the time of admission (except hair loss).
  5. The organ systems of the subjects were as follows:

     1. Diabetes mellitus with poorly controlled blood sugar.
     2. Severe lung disease (Common Terminology Criteria for Adverse Events Version 4.03（CTCAE V4.03）, III-IV).
     3. Active heart disease (Note 3) (New York Heart Association grade III and IV).
     4. Has significant renal or liver dysfunction.
     5. Poorly controlled active hepatitis B or C disease (Note 4).
     6. Primary central nervous system lymphoma or metastasis of central nervous system lymphoma.
     7. A history of mental illness or emotional disorder is judged by a researcher or psychiatrist (Note 5).
  6. Occurrence of disease transformation (such as Richter syndrome, prolymphocytic leukemia, etc.).
  7. Combined use of drugs that cause prolonged QT interval or twisted ventricular tachycardia.
  8. Clinical severe infection with active > CTCAE V4.03 Grade 2; human immunodeficiency virus (HIV) is known to be positive.
  9. Persistent diarrhea (duration ≥ 14 days).
  10. There are other active malignant tumors that may interfere with this study.
  11. Anything that significantly affects the parameters of pharmacokinetics.
  12. Currently receiving moderate and potent cytochrome P450 (CYP) 3A4 isozyme inhibitors or induction drugs (Note 6).
  13. Are participating in other clinical trials.
  14. Any condition that is unstable or may endanger the safety of subjects and their compliance with the study.
  15. The researchers believe that it is not suitable for subjects treated with this regimen.

Note 1: subjects who began to receive erythropoietin or daipotene within 2 weeks before entering the group can be enrolled in the group.

Note 2: if used to treat diseases other than lymphoma, such as rheumatoid arthritis, rheumatic polymyalgia, adrenocortical dysfunction or asthma, subjects can receive a maximum daily dose of 10mg with a stable dose of prednisone.

Note 3: includes any of the following: left ventricular ejection fraction (LVEF) found by cardiac radionuclide scanning (Multigated Radionuclide Angiography (MUGA) ) or echocardiography (ECHO) < 45% Fridericia corrected QT (between QTcF ) > 450ms (QTcF formula); unstable angina pectoris; symptomatic pericarditis; abnormal recording of the left ventricular wall in areas with persistent elevated myocardial enzymes or persistent LVEF function measurements in the past 6 months of myocardial infarction. Has a history of congestive heart failure (New York College of Cardiology Cardiac function Classification III-IV), has a record of cardiomyopathy.

Note 4: a detailed assessment of the history and risk factors of hepatitis B / C must be performed on all subjects during screening. In screening all subjects with positive medical history, quantitative detection of hepatitis B virus deoxyribonucleic acid (DNA) and hepatitis C virus (HCV) ribonucleic acid (RNA) was needed based on risk factors and previous confirmation of hepatitis B/C virus infection. Hepatitis B/C virus replication within the normal range can be included in this study.

Note 5: including medical records of depressive episodes, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, suicidal attempts or suicidal ideation, or thoughts of "causing harm to others immediately", anxiety level 3 or above, etc.

Note 6: allow a combination of inhibitors for weak CYP3A; a list of CYP3A4 inhibitors or inducers is shown in Annex 2 of the study scheme.

* Dose expansion phase:

  1. Severe allergies to research drugs or any of their excipients are known.
  2. Because the research drugs may have genotoxicity, mutagenicity and teratogenicity, the following subjects should be excluded: men and women who plan to reproduce within 5 years without in vitro preservation of sperm or eggs before the trial, unless follow-up studies confirm reproductive safety; pregnant or lactating women.
  3. The treatment of the subjects before the trial:

     1. Before enrolling the group, the subjects had been treated with any persistent or intermittent small molecular targeted drugs (Phosphoinositide 3-kinase (PI3K) inhibitors or Mammalian Target of Rapamycin (mTOR) inhibitors or Histone Deacetylase (HDAC) inhibitors). Subjects in the dose increasing phase of this study will not be subject to the exclusion criteria of this article if they participate in the expanded group phase screening.
     2. Subjects received any hematopoietic colony stimulating factor therapy (such as granulocyte colony stimulating factor （G-CSF）, granulocyte macrophage colony stimulating factor（GM-CSF）) within 2 weeks before enrolling the group (Note 1).
     3. Major surgery was performed within 14 days before enrolling the group, or the side effects of the operation were not stable.
     4. Subjects received glucocorticoid prednisone daily >10mg (or equivalent drug) treatment within 7 days before enrollment. (Note 2)
  4. After the previous treatment (chemotherapy or biotherapy), there was persistent toxicity of grade 2 or above, which was not stable at the time of admission (except hair loss).
  5. The organ systems of the subjects were as follows:

     1. Diabetes mellitus with poorly controlled blood sugar.
     2. Severe lung disease (Common Terminology Criteria for Adverse Events Version 4.03（CTCAE V4.03）, III-IV).
     3. Active heart disease (Note 3) (New York Heart Association grade III and IV).
     4. Has significant renal or liver dysfunction.
     5. Poorly controlled active hepatitis B or C disease (Note 4).
     6. Primary central nervous system lymphoma or metastasis of central nervous system lymphoma.
     7. A history of mental illness or emotional disorder is judged by a researcher or psychiatrist (Note 5).
  6. Occurrence of disease transformation (such as Richter syndrome, prolymphocytic leukemia, etc.).
  7. Combined use of drugs that cause prolonged QT interval or twisted ventricular tachycardia.
  8. Clinical severe infection with active > CTCAE V4.03 Grade 2; human immunodeficiency virus (HIV) is known to be positive.
  9. Persistent diarrhea (duration ≥14 days).
  10. There are other active malignant tumors that may interfere with this study.
  11. Anything that significantly affects the parameters of pharmacokinetics.
  12. Currently receiving moderate and potent cytochrome P450 (CYP) 3A4 isozyme inhibitors or induction drugs (Note 6).
  13. Are participating in other clinical trials.
  14. Any condition that is unstable or may endanger the safety of subjects and their compliance with the study.
  15. The researchers believe that it is not suitable for subjects treated with this regimen.

Note 1: subjects who began to receive erythropoietin or daipotene within 2 weeks before entering the group can be enrolled in the group.

Note 2: if used to treat diseases other than lymphoma, such as rheumatoid arthritis, rheumatic polymyalgia, adrenocortical dysfunction or asthma, subjects can receive a maximum daily dose of 10mg with a stable dose of prednisone.

Note 3: includes any of the following: left ventricular ejection fraction (LVEF) found by cardiac radionuclide scanning (Multigated Radionuclide Angiography (MUGA) ) or echocardiography (ECHO) < 45% Fridericia corrected QT (between QTcF) > 450ms (QTcF formula); unstable angina pectoris; symptomatic pericarditis; abnormal recording of the left ventricular wall in areas with persistent elevated myocardial enzymes or persistent LVEF function measurements in the past 6 months of myocardial infarction. Has a history of congestive heart failure (New York College of Cardiology Cardiac function Classification III-IV), has a record of cardiomyopathy.

Note 4: a detailed assessment of the history and risk factors of hepatitis B / C must be performed on all subjects during screening. In screening all subjects with positive medical history, quantitative detection of hepatitis B virus deoxyribonucleic acid (DNA) and hepatitis C virus (HCV) ribonucleic acid (RNA) was needed based on risk factors and previous confirmation of hepatitis B/C virus infection. Hepatitis B/C virus replication within the normal range can be included in this study.

Note 5: including medical records of depressive episodes, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, suicidal attempts or suicidal ideation, or thoughts of "causing harm to others immediately", anxiety level 3 or above, etc.

Note 6: allow a combination of inhibitors for weak CYP3A; a list of CYP3A4 inhibitors or inducers is shown in Annex 2 of the study scheme.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-03-02 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-03-08 (Actual)

PRIMARY OUTCOMES:
DLT | Dose escalation phase: a 6-day observation after a single administration, cycle 1st of continuous medication (21 days). Dose expansion phase: from date of administration until the date of disease progression or withdrawal, assessed up to 36 months.
  Dose-limiting toxicity
MTD | Dose escalation phase: a 6-day observation after a single administration, cycle 1st of continuous medication (21 days). Dose expansion phase: from date of administration until the date of disease progression or withdrawal, assessed up to 36 months.
  Maximum tolerated dose

SECONDARY OUTCOMES:
AE | From the first administration of the study drug to 30 days after the last administration of the study drug.
  Adverse Event
Cmax | Day 1 and Day 12 of cycle 1 before and within 24 hours after administration (each cycle is 21 days).
  Peak Plasma Concentration
Tmax | Day 1 and Day 12 of cycle 1 before and within 24 hours after administration (each cycle is 21 days).
  Time of peak Plasma Concentration
t1/2 | Day 1 and Day 12 of cycle 1 before and within 24 hours after administration (each cycle is 21 days).
  Half-life of plasma drug concentrations
AUC0-24h | Day 1 and Day 12 of cycle 1 before and within 24 hours after administration (each cycle is 21 days).
  Area under the blood concentration time curve from 0 to 24 hours after administration
AUC0-last | Day 1 and Day 12 of cycle 1 before and within 24 hours after administration (each cycle is 21 days).
  Area under the blood concentration time curve from time zero to the last dose
CL/F | Day 1 and Day 12 of cycle 1 before and within 24 hours after administration (each cycle is 21 days).
  Apparent total plasma clearance
Vd | Day 1 and Day 12 of cycle 1 before and within 24 hours after administration (each cycle is 21 days).
  Apparent volume of distribution
ORR | From date of administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months.
  Objective response rate
DCR | From date of administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months.
  disease control rate
PFS | From date of administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months.
  progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Hui Zhou, Phd, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China